CLINICAL TRIAL: NCT04485468
Title: Integrated Parkinson Care Networks: Assessment of Economics and Socials Barriers to the Optimal Care Pathway for Parkinson Disease Patients
Brief Title: Integrated Parkinson Care Networks: Assessment of Economics and Socials Barriers
Acronym: ECOSO-ICAREPD
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0184
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease,; Socio-economic
MeSH Terms: conditions — Parkinson Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's disease patients: Parkinson's disease patients and over 18 years old
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The patient answers the questionnaire directly following his consultation or teleconsultation or may arrange a telephone appointment with the clinical research associate a little later.

SUMMARY:
According to the latest public health report in France, Parkinson's disease (PD) affects around 160,000 patients.

It is therefore essential to estimate the overall consumption of medical and non-medical resources by patients with PD in order to characterize the share of medical and non-medical care reimbursed by health insurance, the share of medical and non-medical care not reimbursed. by health insurance, as well as the share of formal and informal care in order to identify potential economic barriers to an optimal care path for patients with PD. It is also necessary to have information on the socio-economic characteristics and the place of residence of the resident in order to estimate the impact of these determinants on an optimal course of care.

DETAILED DESCRIPTION:
According to the latest public health report in France, Parkinson's disease (PD) affects around 160,000 patients

The coordination of the care pathway for patients with Parkinson disease has been improved since the implementation on the national territory of 7 interregional coordination centers and 25 regional expert centers in 2012.

Health insurance reimburses 100% of direct medical and non-medical care as soon as patients are registered in Long-Term Condition n°16. However, we currently have little information about care that is not recognized for financial coverage by health insurance.

It is therefore essential to estimate the overall consumption of medical and non-medical resources by patients with PD in order to characterize the share of medical and non-medical care reimbursed by health insurance, the share of medical and non-medical care not reimbursed. by health insurance, as well as the share of formal and informal care in order to identify potential economic barriers to an optimal care path for patients with PD. It is also necessary to have information on the socio-economic characteristics and the place of residence of the resident in order to estimate the impact of these determinants on an optimal course of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease of any stage of severity
* Patients over 18 years of age
* Patients living at home
* Patient consultant at the expert center Parkinson's at Toulouse University Hospital

Exclusion Criteria:

* Pregnant and lactating woman
* Patient under guardianship, curatorship or safeguard of justice
* Person who does not understand French to be able to answer the questionnaire
* Patient who participated or participated in the iCare PD project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease patients and over 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Identify the economic barriers to an optimal care path | Day 0
  It is the collection of the number of resources consumed and the remainder to be borne by the patient as well as the number of hours of informal help that will be valued using the replacement cost approach.

SECONDARY OUTCOMES:
Identify and quantify the cost of the care pathway for patients with Parkinson's disease | Day 0
  it is the quantification of the number of resources consumed and identification of the unit costs for each type of resources consumed.
identify socio-economic determinants | Day 0
  identify the socio-economic and territorial determinants that could have an impact on an optimal care path.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Rascol, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No